CLINICAL TRIAL: NCT02405676
Title: Treatment Regimen or Children or Adolescent with Mature B-cell NHL or B-AL in China
Brief Title: BNHL-2015 for Children or Adolescents in China
Acronym: BNHL-2015
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Children's Cancer Group, China (Network)
Collaborators: Tongji Hospital (Other); Nanjing Children's Hospital (Other); West China Second University Hospital (Other); Xiangya Hospital of Central South University (Other); Qilu Hospital of Shandong University (Other); Children's Hospital of Soochow University (Other); Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Yi-Jin Gao, Shanghai Children's Medical Center, School of Medicine, Shanghai Jiaotong University, Shanghai, China, Children's Cancer Group, China
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCCG-BNHL-2015
Record Dates: First submitted 2015-02-26; First posted 2015-04-01 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Mature B-cell Non-Hodgkin Lymphoma
Keywords: Lymphoma; non-Hodgkin; B-lymphocytes; Child; Multicenter study
MeSH Terms: conditions — Lymphoma | interventions — Prednisone; Vincristine; Cyclophosphamide; Cytarabine; Etoposide; Methotrexate; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Risk group 1 (Other): Complete resection of stage I or II disease: 3 courses (A-B-A) and 3 intrathecal injections(Cytarabine/Methotrexate/Dexamethasone, age adjusted);
  Interventions: Drug: Cyclophosphamide, Vincristine, Cytarabine, Doxorubincin, Prednisone; Drug: Ifosphamide, Etoposide, Methotrexate, Vincristine, Prednisone
- Risk group2 (Other): Not or incompletely resected stage I/II disease and LDH <2 times NL: 5 courses (A--B--A--B--A) and 8 intrathecal injections;
  Interventions: Drug: Cyclophosphamide, Vincristine, Cytarabine, Doxorubincin, Prednisone; Drug: Ifosphamide, Etoposide, Methotrexate, Vincristine, Prednisone
- Risk group3 (Other): Stage III with high LDH < 4 times NL, or Stage I,II with LDH >=2 times NL: Preface followed by 6 courses (P(Cyclophosphamide/Vincristine/Prednisone)-A-BB-AA-BB-AA-BB) and 13 intrathecal injections; Dosage of Cytarabine, Methotrexate and Etoposide was increased in AA or BB compared with A or B. Vindelsine was used in AA/BB instead of Vincristine in A/B.
  Interventions: Drug: Prednisone,Vincristine, Cyclophosphamide; Drug: Cyclophosphamide, Vincristine, Cytarabine, Doxorubincin, Prednisone; Drug: Cyclophosphamide, Vindelsine, Cytarabine, Doxorubincin, Prednisone; Drug: Ifosphamide, Etoposide, Methotrexate, Vindelsine, Prednisone
- Risk group4 (Other): Stage III with LDH≥4N, or Stage IV, or B-AL: Preface followed by 4 dose of rituximab (375mg/m2) combined 6 courses of chemotherapy, together with 13 intrathecal injections: P-A-(Rituximab)BB-(Rituximab)AA-(Rituximab)BB-(Rituximab)AA-BB; rituximab is at D0 of each course.
  Interventions: Drug: Prednisone,Vincristine, Cyclophosphamide; Drug: Cyclophosphamide, Vincristine, Cytarabine, Doxorubincin, Prednisone; Drug: Cyclophosphamide, Vindelsine, Cytarabine, Doxorubincin, Prednisone; Drug: Ifosphamide, Etoposide, Methotrexate, Vindelsine, Prednisone; Drug: Rituximab

INTERVENTIONS:
Drug: Prednisone,Vincristine, Cyclophosphamide — Prednisone 45mg/m2, D1~7; Vincristine 1.5mg/m2(MAX 2mg), D1; Cyclophosphamide 300mg/m2, D1; Intrathecal injection, D1;
  Other Names: Preface
  Arms: Risk group3; Risk group4
Drug: Cyclophosphamide, Vincristine, Cytarabine, Doxorubincin, Prednisone — Cyclophosphamide 800mg/m2, D1, then 200mg/m2, D2~4;Vincristine 1.5mg/m2 (MAX 2mg), D1; Cytarabine 1g/m2/dose, (2 doses, 12-hour interval), D4;Doxorubincin 20mg/m2, D2,3; Prednisone 60mg/m2, D1~7;Intrathecal injection, D1,8;
  Other Names: Protocol A
Drug: Ifosphamide, Etoposide, Methotrexate, Vincristine, Prednisone — Ifosphamide 1.2g/m2, D1~5; Etoposide, 60mg/m2, D3~5; Methotrexate, 0.5g/m2, D1;Vincristine 1.5mg/m2 (MAX 2mg), D1; Prednisone 60mg/m2, D1~7;Intrathecal injection, D1;
  Other Names: Protocol B
  Arms: Risk group 1; Risk group2
Drug: Cyclophosphamide, Vindelsine, Cytarabine, Doxorubincin, Prednisone — Cyclophosphamide 800mg/m2, D1, then 200mg/m2, D2~4;Vindelsine 3mg/m2 (MAX 5mg), D1; Cytarabine 2g/m2/dose, (2 doses, 12-hour interval), D4;Doxorubincin 20mg/m2, D2,3; Prednisone 60mg/m2, D1~7;Intrathecal injection, D1,8;
  Other Names: Protocol AA
  Arms: Risk group3; Risk group4
Drug: Ifosphamide, Etoposide, Methotrexate, Vindelsine, Prednisone — Ifosphamide 1.2g/m2, D1~5; Etoposide, 100mg/m2, D3~5; Methotrexate, 5g/m2, D1;Vindelsine 3mg/m2 (MAX 5mg), D1; Prednisone 60mg/m2, D1~7;Intrathecal injection, D1,8;
  Other Names: Protocol BB
  Arms: Risk group3; Risk group4
Drug: Rituximab — 375mg/m2, 4 injections for patients in Risk group4; D0 of Protocol AA or BB;
  Arms: Risk group4

SUMMARY:
The purpose of this study is to test whether adding 4 injections of rituximab and increasing the intensity of chemotherapy regimens in advanced patients can improve the EFS compared with the historical study CCCG-NHL-2010.

DETAILED DESCRIPTION:
In our previous study (CCCG-NHL-2010), two-year EFS was 100% for Stage I, 91.3% ± 6.1% for Stage II, 75.8% ± 4.4% for Stage III, 56.3% ± 13.5% for Stage IV, and 36.4% ± 14.5% for B-AL, respectively. To improve survival for pediatric patients with B-NHL/B-AL, the investigators launched a new study in China. Compared with our previous treatment regimens (CCCG-2010), patients with stage III and LDH>4 times NL, any stage IV or B-AL were stratified into R4. The dose of methotrexate was increased to 5000mg/m2 for patients in R3 or R4 (previously 3000mg/m2). Four injections of rituximab was added to the chemotherapy for patients in R4. Our aim is to test whether adding rituximab or high dose of methotrexate (5000mg/m2) would improving 2-year EFS for patients in advanced groups.

ELIGIBILITY:
Inclusion Criteria:

* Histology or cytologically confirmed matureB-cell NHL/AL(Burkitt, DLBCL, PMLBL,or aggressive mature B-cell NHL non other specified or specifiable)
* Able to comply with scheduled follow-up and with management of toxicity
* Signed informed consent

Exclusion Criteria:

* Follicular lymphoma, MALT and nodular marginal zone are not included into this therapeutic study
* Patients with congenital immunodeficiency, chromosomal breakage syndrome, prior organ transplantation, previous malignancy of any type, or known positive HIV serology.
* -Evidence of pregnancy or lactation period.

  * Past or current anti-cancer treatment except corticosteroids during less than one week.

Exclusion criteria related to rituximab:

* Tumor cell negative for CD20.
* Prior exposure to rituximab.
* Hepatitis B carrier status history of HBV or positive serology.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2015-01; Primary Completion 2023-12-31 (Actual); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 2 year

SECONDARY OUTCOMES:
Overall survival | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Jin Gao, MD, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- West China Second University Hospital of Sichuan University, Chengdu, Sichuan, China

REFERENCES:
- [Background] Reiter A, Schrappe M, Tiemann M, Ludwig WD, Yakisan E, Zimmermann M, Mann G, Chott A, Ebell W, Klingebiel T, Graf N, Kremens B, Muller-Weihrich S, Pluss HJ, Zintl F, Henze G, Riehm H. Improved treatment results in childhood B-cell neoplasms with tailored intensification of therapy: A report of the Berlin-Frankfurt-Munster Group Trial NHL-BFM 90. Blood. 1999 Nov 15;94(10):3294-306. PMID 10552938
- [Background] Miles RR, Arnold S, Cairo MS. Risk factors and treatment of childhood and adolescent Burkitt lymphoma/leukaemia. Br J Haematol. 2012 Mar;156(6):730-43. doi: 10.1111/j.1365-2141.2011.09024.x. Epub 2012 Jan 20. PMID 22260323
- [Background] Woessmann W, Seidemann K, Mann G, Zimmermann M, Burkhardt B, Oschlies I, Ludwig WD, Klingebiel T, Graf N, Gruhn B, Juergens H, Niggli F, Parwaresch R, Gadner H, Riehm H, Schrappe M, Reiter A; BFM Group. The impact of the methotrexate administration schedule and dose in the treatment of children and adolescents with B-cell neoplasms: a report of the BFM Group Study NHL-BFM95. Blood. 2005 Feb 1;105(3):948-58. doi: 10.1182/blood-2004-03-0973. Epub 2004 Oct 14. PMID 15486066
- [Background] Meinhardt A, Burkhardt B, Zimmermann M, Borkhardt A, Kontny U, Klingebiel T, Berthold F, Janka-Schaub G, Klein C, Kabickova E, Klapper W, Attarbaschi A, Schrappe M, Reiter A; Berlin-Frankfurt-Munster group. Phase II window study on rituximab in newly diagnosed pediatric mature B-cell non-Hodgkin's lymphoma and Burkitt leukemia. J Clin Oncol. 2010 Jul 1;28(19):3115-21. doi: 10.1200/JCO.2009.26.6791. Epub 2010 Jun 1. PMID 20516455
- [Background] Goldman S, Smith L, Anderson JR, Perkins S, Harrison L, Geyer MB, Gross TG, Weinstein H, Bergeron S, Shiramizu B, Sanger W, Barth M, Zhi J, Cairo MS. Rituximab and FAB/LMB 96 chemotherapy in children with Stage III/IV B-cell non-Hodgkin lymphoma: a Children's Oncology Group report. Leukemia. 2013 Apr;27(5):1174-7. doi: 10.1038/leu.2012.255. Epub 2012 Sep 3. No abstract available. PMID 22940833
- [Derived] Gao YJ, Fang YJ, Gao J, Yan J, Yang LC, Liu AG, Ju XL, Lu J, Han YL, Wang J, Xie M, Guo X, Tang JY. A prospective multicenter study investigating rituximab combined with intensive chemotherapy in newly diagnosed pediatric patients with aggressive mature B cell non-Hodgkin lymphoma (CCCG-BNHL-2015): a report from the Chinese Children's Cancer Group. Ann Hematol. 2022 Sep;101(9):2035-2043. doi: 10.1007/s00277-022-04904-w. Epub 2022 Jul 13. PMID 35829780